CLINICAL TRIAL: NCT06000917
Title: A Multicenter, Single-arm, Prospective Study of Neoadjuvant Pyrotinib Combined With Trastuzumab，Carboplatin and Paclitaxel for ER+/HER2+ Early or Locally Advanced Breast Cancer
Brief Title: A Study of Neoadjuvant TCHpy（Pyrotinib ，Trastuzumab，Carboplatin and Paclitaxel）for ER+/HER2+ Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHCT22745
Record Dates: First submitted 2023-08-08; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer; Neoadjuvant
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pyrotinib,Trastuzumab，carboplatin，Albumin paclitaxel (Experimental): Pyrotinib tablets: 320mg qd, 21 days for 1 cycle, continuous administration of 6 cycles.
  Trastuzumab: The first cycle was 8mg/kg, the second to sixth cycle was 6mg/kg, 21 days was 1 cycle, continuous administration of 6 cycles.
  Albuminpaclitaxel: On the first day of cycle 1, 260mg/m2 was given intravenously, 21 days for 1 cycle, and 6 consecutive cycles were given.
  Carboplatin: Endogenous creatinine clearance was calculated using the Cockcroft formula, with AUC 5 for the 1st to 6th cycle and 1 cycle for the 21st day and 6 consecutive cycles of administration
  Interventions: Drug: pyrotinib,Trastuzumab，carboplatin，Albumin paclitaxel

INTERVENTIONS:
Drug: pyrotinib,Trastuzumab，carboplatin，Albumin paclitaxel — Pyrotinib tablets: 320mg qd, oral administration after breakfast, 21 days for 1 cycle, continuous administration of 6 cycles.
  Trastuzumab: The first cycle was 8mg/kg, the second to sixth cycle was 6mg/kg, 21 days was 1 cycle, continuous administration of 6 cycles.
  Albuminpaclitaxel: On the first day of cycle 1, 260mg/m2 was given intravenously, 21 days for 1 cycle, and 6 consecutive cycles were given.
  Carboplatin: Endogenous creatinine clearance was calculated using the Cockcroft formula, with AUC 5 for the 1st to 6th cycle and 1 cycle for the 21st day and 6 consecutive cycles of administration

SUMMARY:
This study is a multicenter, single-arm, prospective, open clinical study to evaluate the efficacy and safety of pyrotinib in combination with trastuzumab, albumin paclitaxel, and carboplatin in neoadjuvant therapy for ER+/HER2+ early or locally advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Newly treated female patients aged ≥18 years and ≤75 years;
* ECOG score 0~1;
* Pathologically diagnosed as HER2-positive breast cancer patients with early or locally advanced tumor stage, primary tumor diameter T≥2cm or lymph node positive;
* Hormone receptor status (ER and PgR) is known, where ER≥10%
* Normal function of major organs:

  1. The standard of blood routine examination should meet: ANC ≥1.5×109/L; PLT≥90×109/L; Hb ≥90g/L
  2. Biochemical examination should meet the following standards: TBIL≤ the upper limit of normal value(ULN); ALT and AST≤1.5 times the upper limit of normal (ULN); Alkaline phosphatase ≤2.5 times the upper limit of normal (ULN); BUN and Cr≤1.5×ULN and creatinine clearance ≥50 mL/min (CockcroftGault formula);
  3. Cardiac color ultrasound and echocardiography: left ventricular ejection fraction(LVEF≥55%)
  4. Fridericia calibrated QT interval (QTcF) for 18-lead ECG <470 ms;
* For female patients who are not menopausal or have not been surgically sterilized: consent to abstinence or use of an effective contraceptive method during treatment and for at least 7 months after the last dose in the study treatment;
* Volunteer to join the study and sign the informed consent.

Exclusion Criteria:

* Stage IV (metastatic) breast cancer;
* Inflammatory breast cancer;
* Previous antitumor therapy or radiation therapy for any malignancies, excluding cured cervical carcinoma in situ, basal cell carcinoma, or squamous cell carcinoma;
* Also receiving antitumor therapy in other clinical trials, including endocrine therapy, bisphosphonate therapy, or immunotherapy;
* Had a major surgery not related to breast cancer in the 4 weeks prior to enrollment, or had not fully recovered from such surgery;
* Serious heart disease or discomfort, including but not limited to the following:

  * History of heart failure or systolic dysfunction (LVEF < 50%)
  * High-risk uncontrolled arrhythmias, such as atrial tachycardia, resting heart rate >100 bpm, significant ventricular arrhythmias (such as ventricular tachycardia), or higher-grade atrioventricular block (i.e. Mobitz II second- degree atrioventricular block or third-degree atrioventricular block
* Inability to swallow, intestinal obstruction, or other factors affecting the use and absorption of the drug;
* Known allergic history of the drug components of this protocol; A history of immunodeficiency, including HIV testing positive, or other acquired, congenital immunodeficiency diseases, or a history of organ transplantation;
* Women who are pregnant or nursing, women who are fertile and have a positive baseline pregnancy test, or women of childbearing age who are unwilling to use effective contraception throughout the trial period and within 7 months after the last study medication;
* Have a serious concomitant condition or other comorbid condition that interferes with planned treatment, or any other condition in which the investigator deems the patient unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2025-05-11 (Estimated); Study Completion 2028-05-11 (Estimated)

PRIMARY OUTCOMES:
total Pathological Complete Response(tPCR) | 2 years

SECONDARY OUTCOMES:
breast Pathological Complete Response(bPCR) | 2 years
overall response rate(ORR) | 2 years
event-free survival(EFS) | 5 years

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - WuhanHU, Wuhan, Hubei
  - Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No